CLINICAL TRIAL: NCT05543499
Title: Database: Standardized Prenatal Management and Perinatal Outcome of Complicated Monochorionic Pregnancies
Brief Title: Database of Monochorionic Pregnancies
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Rodrigo Ruano, Professor and Chief of MFM Division, University of Miami
Other Study IDs: 20210709
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Monochorionic Diamniotic Placenta; Monochorial Monoamniotic Placenta; Twin; Complicating Pregnancy; Twin to Twin Transfusion Syndrome; Twin Reversal Arterial Perfusion Syndrome
Keywords: multiple pregnancies; Twins
MeSH Terms: conditions — Pregnancy Complications; Fetofetal Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Monochorionic Pregnancy Group: Participants with complicated monochorionic pregnancies (MC) will be followed prospectively beginning at the time of the mother's evaluation for a complication related to monochorionic (MC) multiple pregnancies through delivery of the child and follow-up of the child to 12 months of life.

SUMMARY:
The purpose of this study is to collect and analyze data regarding natural history, indications for fetal interventions, and maternal and fetal/neonatal outcomes associated with complicated monochorionic twin pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of MC pregnancies (maternal, fetal, and neonatal data) that have undergone evaluation and/or treatment for complications attributable to monochorionic twin pregnancy at the University of Miami.
* Maternal age 18 years and older.

Exclusion Criteria:

* Participation declined or consent not granted in prospective arm
* Loss to follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of Monochorionic pregnancies (maternal, fetal, and neonatal data) that have undergone evaluation and/or treatment for complications attributable to monochorionic twin pregnancy at the University of Miami.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Preterm Delivery | Up to 42 weeks gestation
  Preterm delivery is defined as birth <37 weeks gestation
Number of participant with Premature Spontaneous Rupture of the Membranes | Up to 42 weeks
  As per clinical evaluation
Number of Infant Deaths | Up to 12 months post infant delivery
  The Number of Infant Deaths

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ruano, MD PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No